CLINICAL TRIAL: NCT00706602
Title: International Collaborative Effort on Chronic Obstructive Lung Disease: Exacerbation Risk Index Cohorts
Brief Title: Predicting the Course of Chronic Obstructive Pulmonary Disease (COPD) in Primary Care
Acronym: ICECOLDERIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Zurich Lung League (Other); The Netherlands Asthma Foundation (Other)
Responsible Party: Milo A Puhan/MD PhD, University of Zurich and Johns Hopkins University
Other Study IDs: 3233B0-115216; 3.4.07.045
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: COPD
Keywords: COPD; prognosis; prediction rule; health-related quality of life; risk factors; derivation; validation; exacerbation; mortality; primary care; treatment; decision making
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Swiss COPD cohort
- 2: Dutch COPD cohort

SUMMARY:
Background: COPD is a systemic illness; morbidity and mortality due to this disease are on the increase, and it has great impact on patients' lives. Most COPD patients are managed by general practitioners (GP). GPs base their initial assessment of patients' disease severity mainly on lung function and then inform patients about adequate treatment. However, lung function correlates poorly with COPD-specific health-related quality of life and exacerbation frequency. Preventive cardiology embraced risk index-guided treatment successfully. COPD disease severity indices that better represent the clinical manifestations of COPD are needed that can be used to guide risk-stratified treatment.

Objectives: (1) The development and validation of a practical COPD disease severity index to predict the course of health-related quality of life over time. (2) The validation of the ADO-Index (Age, Dyspnea, Obstruction) to predict 3-year mortality in COPD patients in primary care. (3) Link evidence on treatment effects to the COPD risk indices to guide COPD treatment selection.

Methods: We are in the process of conducting two linked prospective cohort studies with 413 COPD patients (GOLD stages 2-4) from GPs in Switzerland and the Netherlands. We performed a sound baseline assessment including detailed patient history, lung function, measurement of exercise capacity and blood sampling. During the follow-up of at least five years, we update the patients' profile by registering health status, exacerbations and health-related quality of life and, after 2 years, lung function and measurement of exercise capacity. For aim 1, we will identify the best combination of variables predicting the course of health-related quality of life over time using multivariable regression analysis. For aim 2, we will assess discrimination and calibration of the ADO index to predict 3-year mortality. For aim 3, we will estimate treatment effects for individual patient profiles using complex statistical models such as Markov models.

Significance of project: After this study, different risk scores will be available for use in primary care so that general practitioners can estimate what impact COPD will have on the patients. By linking these risk scores to evidence form treatment studies, it will be possible to show for an individual patient how COPD and different treatments impacts on mortality, symptoms and exacerbations. Thereby, patients and physicians can make more informed treatment decisions balancing the benefits and downsides of different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥40 years of age with COPD in GOLD stage II to IV (postbronchodilator FEV1/FVC≤0.70, postbronchodilator FEV1≤80% predicted) are eligible if in- or outpatient treatment of their last exacerbation ended ≥4 weeks ago.

Exclusion Criteria:

* Patients who received mechanical ventilation in the previous 12 months (because of extremely poor prognosis), patients with co-morbidities associated with a life expectancy of ≤12 months, patients diagnosed with dementia, psychosis or other psychiatric illness that invalidate assessment of patient-reported parameters and patients who cannot complete thr baseline assessment due to language difficulties.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients from primary care. Patients are identified through electronic or paper-based patient charts and by participating general practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Chronic Respiratory Questionnaire | At least 5 years

SECONDARY OUTCOMES:
Exacerbation | At least 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Milo A Puhan, MD PhD, Principal Investigator — University of Zurich, Switzerland
Locations (1):
- Institute for primary care, University of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Siebeling L, ter Riet G, van der Wal WM, Geskus RB, Zoller M, Muggensturm P, Joleska I, Puhan MA. ICE COLD ERIC--International collaborative effort on chronic obstructive lung disease: exacerbation risk index cohorts--study protocol for an international COPD cohort study. BMC Pulm Med. 2009 May 6;9:15. doi: 10.1186/1471-2466-9-15. PMID 19419546
- [Derived] Tai AS, Liao LH, Lin SH. On the Conventional Definition of Path-specific Effects: Fully Mediated Interaction With Multiple Ordered Mediators. Epidemiology. 2022 Nov 1;33(6):817-827. doi: 10.1097/EDE.0000000000001520. Epub 2022 Jun 24. PMID 36220579
- [Derived] Steurer-Stey C, Dalla Lana K, Braun J, Ter Riet G, Puhan MA. Effects of the "Living well with COPD" intervention in primary care: a comparative study. Eur Respir J. 2018 Jan 4;51(1):1701375. doi: 10.1183/13993003.01375-2017. Print 2018 Jan. PMID 29301921
- [Derived] Strassmann A, Frei A, Haile SR, Ter Riet G, Puhan MA. Commonly Used Patient-Reported Outcomes Do Not Improve Prediction of COPD Exacerbations: A Multicenter 4(1/2) Year Prospective Cohort Study. Chest. 2017 Dec;152(6):1179-1187. doi: 10.1016/j.chest.2017.09.003. Epub 2017 Sep 18. PMID 28923760
- [Derived] Crook S, Frei A, Ter Riet G, Puhan MA. Prediction of long-term clinical outcomes using simple functional exercise performance tests in patients with COPD: a 5-year prospective cohort study. Respir Res. 2017 Jun 2;18(1):112. doi: 10.1186/s12931-017-0598-6. PMID 28578705
- [Derived] Frei A, Siebeling L, Wolters C, Held L, Muggensturm P, Strassmann A, Zoller M, Ter Riet G, Puhan MA. The Inaccuracy of Patient Recall for COPD Exacerbation Rate Estimation and Its Implications: Results from Central Adjudication. Chest. 2016 Oct;150(4):860-868. doi: 10.1016/j.chest.2016.06.031. Epub 2016 Aug 26. PMID 27400907
- [Derived] Frei A, Muggensturm P, Putcha N, Siebeling L, Zoller M, Boyd CM, ter Riet G, Puhan MA. Five comorbidities reflected the health status in patients with chronic obstructive pulmonary disease: the newly developed COMCOLD index. J Clin Epidemiol. 2014 Aug;67(8):904-11. doi: 10.1016/j.jclinepi.2014.03.005. Epub 2014 Apr 29. PMID 24786594
- [Derived] Puhan MA, Siebeling L, Frei A, Zoller M, Bischoff-Ferrari H, Ter Riet G. No association of 25-hydroxyvitamin D with exacerbations in primary care patients with COPD. Chest. 2014 Jan;145(1):37-43. doi: 10.1378/chest.13-1296. PMID 24008868
- [Derived] Puhan MA, Siebeling L, Zoller M, Muggensturm P, ter Riet G. Simple functional performance tests and mortality in COPD. Eur Respir J. 2013 Oct;42(4):956-63. doi: 10.1183/09031936.00131612. Epub 2013 Mar 21. PMID 23520321